CLINICAL TRIAL: NCT03049397
Title: Family Functioning and Bereavement Outcomes Following the Enhancing Connections Program in Palliative Care
Brief Title: Enhancing Connections Program in Improving Family Adjustment in Patients With Incurable Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Pilot deemed not feasible based on predetermined stopping rules
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9667; NCI-2016-01640 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9667 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9218011 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Advanced Malignant Neoplasm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Enhancing Connections program) (Experimental): Patients and co-parents participate in the Enhancing Connections program consisting of 5 sessions over 1 hour each in the clinic or over the telephone. Session topics include managing cancer-related emotions when talking to children, developing deep listening skills, initiating difficult cancer-related conversations with children, interpreting a child's behavior, recognizing newly acquired gains from the program, and identifying available resources that can be used after program completion.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Communication Intervention — Complete Enhancing Connections program
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well the Enhancing Connections program improves family adjustment in patients with incurable cancer. Participating in an educational program with a co-parent to learn about ways to talk to a child about cancer may help parents and co-parents support their child with the parent's cancer and may help families communicate and function better.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility of the study protocol in advanced cancer patients and co-parents (recruitment/retention, dosage and fidelity of the intervention; program acceptability of program; and logistics).

II. Evaluate the short-term impact of the program on the diagnosed parents', co-parents' and children's adjustment and family functioning using a within group design (pre- and posttest design).

III. Compare outcomes from the Enhancing Connections Palliative Program with similar outcomes obtained from the completed phase III trial (between group design) for the patients and children outcomes.

IV. Evaluate the longer term impact of the program on the co-parents' and children's adjustment, including bereavement outcomes when appropriate, using a within and across group design (pre- and posttest design).

OUTLINE:

Patients and co-parents participate in the Enhancing Connections program consisting of 5 sessions over 1 hour each in the clinic or over the telephone. Session topics include managing cancer-related emotions when talking to children, developing deep listening skills, initiating difficult cancer-related conversations with children, interpreting a child's behavior, recognizing newly acquired gains from the program, and identifying available resources that can be used after program completion.

After completion of the study, participants are followed-up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* Ages 25-65 years
* Have a diagnosis of incurable cancer of any type; at any time in the diagnosis as long as they have at least a 4 month life expectancy based on the opinion of the attending physician
* Read and write English among their languages of choice
* Parent must live at least 50% of the time in the home and have a child 5-17 years old living at home who has been told their parent's cancer diagnosis

CO-PARENTS

* Co-parents must reside with the consenting eligible cancer participant (and child) at least 50% of the time and be actively participating in the care of the child
* If a biological parent lives in the home, and is physically well themselves, this person must be the co-parent
* If a biological parent does not live in the home (or has died), the co-parent does not have to be a biological parent; therefore, co-parents may be step-parents, lesbian, gay, bi-sexual or transgender (LGBT) partners, grandparents, aunts, uncles, etc if they otherwise meet eligibility criteria
* He or she can read and write English among their languages of choice and agrees to attend the patient intervention sessions in person or by telephone

CHILDREN

* The patient and co-parent must agree to focus on the same child throughout the study and consent to have the child participate before the child's assent will be sought
* Children aged 5-13 years of age will participate with a waiver of assent
* Children aged 14-17 will assent to participate in the research study by signing a separate assent form
* Children of formal assenting age will be eligible to participate if they can read and write English among their languages of choice

ALL PARTICIPANTS

* Participants must live within 35 miles of the University of Washington, Seattle, WA to receive the in-person version of the intervention
* Parents and co-parents selecting the telephone version of the intervention may live any distance from the University of Washington

Exclusion Criteria:

* Patients will be excluded if they are enrolled in hospice at time of enrollment; however, they will be allowed to continue in the study if they enroll in hospice after beginning the study
* The triad will be ineligible if any member lives in the home less than 50% of the time
* If any member of the triad retracts consent or assent prior to completion of the post-intervention surveys, then all members will be excluded from the study thereafter
* The child will be excluded if he or she has learning challenges as assessed by the patient or co-parent; patients and co-parents will be instructed to consider any formal diagnoses of a learning disability of the presence of an Individual Education Plan (IEP) when making this assessment

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Enhancing Connections program in advanced cancer patients and co-parents | Up to 2 years
  Recruitment and retention of all triads will be monitored. Dosage and fidelity will be monitored for each intervention session. Program acceptability (per session, overall, duration of program, interval between intervention sessions) will be assessed from a debriefing interview. For logistics four areas will be monitored: rate of receipt of mailed materials both to participants and from participants; duration and type (whether telephone or in-person) of intervention sessions; rate of success in scheduling and completing intervention sessions with patient and co-parent; and quality of data on baseline, post-intervention and follow-up measures.
Change in adjustment and family functioning | Baseline to 6 months
  Descriptive statistics (e.g. means, medians) will be used to describe the Enhancing Connections palliative care population. Parents', co-parents and children's baseline scores [parent-reported] on standardized questionnaires will be compared with post-intervention and 6 month follow-up scores on the same measures.
Outcomes from the Enhancing Connections Palliative Program as measured by the Child Behavior Check List | Up to 2 years
  Linear mixed modeling based on Maximum Likelihood Estimation will be used to test the differences between the Child Behavior Check List results for the Enhancing Connections Palliative Program and the completed phase III trial (EC-R01).
Change in adjustment as measured by post-traumatic growth scores | Baseline to 6 months
  Enhancing Connection Palliative Program parents', co-parents' and children's post-traumatic growth scores will be compared with follow-up (6 month) scores on the same measure.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Loggers, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States